CLINICAL TRIAL: NCT05712811
Title: Cryotherapy Versus Topical Tricholoacetic Acid 90% in Treatment of Common Warts
Brief Title: Comparison of Cryotherapy and Peeling Agent in the Treatment of Common Warts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Combined Military Hospital Abbottabad (Other)
Responsible Party: Principal Investigator, Dr kiran gul, Principal investigator, Combined Military Hospital Abbottabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMHAbbottabad
Record Dates: First submitted 2023-01-18; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Warts
MeSH Terms: conditions — Warts | interventions — Cryotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A cryotherapy (Active Comparator): Cryotherapy Group A had their warts treated once every two weeks for a total of twelve weeks, with liquid nitrogen using cryoget method for 10 to 15 seconds on each lesion (depending on size, until a narrow white rim of around 1 mm developed around it).
  Interventions: Drug: CRYOTHERAPY
- Group B Topical TCA 90% (Active Comparator): Topical TCA 90 % Warts in Group B were treated with liquid TCA 90% by an applicator every two weeks for a total of twelve weeks. After 20 minutes, patients were instructed to remove the solution by washing their warts with water or regular saline
  Interventions: Drug: Tricholoracetic acid

INTERVENTIONS:
Drug: CRYOTHERAPY — Group A had their warts treated once every two weeks for a total of twelve weeks, with liquid nitrogen using cryoget method for 10 to 15 seconds on each lesion (depending on size, until a narrow white rim of around 1 mm developed around it).
  Other Names: Liquid nitrogen
  Arms: Group A cryotherapy
Drug: Tricholoracetic acid — Group B were treated with liquid TCA 90% by an applicator every two weeks for a total of twelve weeks. After 20 minutes, patients were instructed to remove the solution by washing their warts with water or regular saline.
  Other Names: Peeling agent
  Arms: Group B Topical TCA 90%

SUMMARY:
Objective: To compare the efficacy of cryotherapy using liquid nitrogen (cryoget method) versus trichloroacetic acid 90% (applicator method) in treatment of common warts.

Study Design: Randomized Control Trial. Place And Duration of Study: Department of Dermatology, CMH Abbottabad from Jun 2022 to Nov, 2022.

DETAILED DESCRIPTION:
A total of 60 patients were enrolled in this investigation by non-probability consecutive sampling technique. Sample size was calculated using WHO sample size calculator and patients were randomized into two equal groups, A and B, each comprising of 30 patients through lottery method. Patients with common warts such as hard lesions, raised lumps with rough surfaces at the back of their fingers, around nails and palm of their hands between the ages of 18 and 60 were included, whereas those with genital warts, cardiac, hepatic, renal, or hypercholesterolemia were excluded.

ELIGIBILITY:
Inclusion Criteria:

* Patient presented with common warts in dermatology opd

Exclusion Criteria:

* • Patients with warts on toes and tip of fingers

  * genital warts
  * cardiac, hepatic and renal disease
  * hypercholesterolemia
  * hypersensitivity reactions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Comparison of cryotherapy and Tricholoracetic acid 90% in treatment of common warts | 12 weeks
  Outcome was determined at the end of third month and the patients were labelled as cured and the efficacy was labelled as "Yes" in cases with absence of all the lesions. After twelve weeks of therapy, individuals with persistent warts were regarded as cases of treatment failure and efficacy was labelled as "No".

CONTACTS AND LOCATIONS:
Locations (1):
- Cmh abbottabad, Abbottābād, Kpk, Pakistan